CLINICAL TRIAL: NCT05711589
Title: Safety and Efficacy of Intracardiac Echocardiography-guided Zero-fluoroscopic Cryoballoon Ablation for Atrial Fibrillation : A Prospective Randomized Controlled Trial
Brief Title: Zero-fluoroscopic Cryoballoon Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HALLYM 2019-04-025-001
Record Dates: First submitted 2023-01-18; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation Paroxysmal
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: zero-fluoroscopic and conventional fluoroscopy groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Placebo Comparator): cryoablation (CBA) was performed under fluoroscopic guidance
  Interventions: Procedure: cryoablation (CBA) was performed under fluoroscopic guidance
- Zero-X group (Experimental): CBA was performed under intracardiac echocardiography guidance without fluoroscopy
  Interventions: Procedure: CBA was performed under intracardiac echocardiography guidance without fluoroscopy

INTERVENTIONS:
Procedure: CBA was performed under intracardiac echocardiography guidance without fluoroscopy — Zero-X group: Patients undergoing ICE-guided CBA
  Arms: Zero-X group
Procedure: cryoablation (CBA) was performed under fluoroscopic guidance — cryoablation (CBA) was performed under fluoroscopic guidance
  Arms: conventional group

SUMMARY:
This study aimed to investigate safety and efficacy of intracardiac echocardiography (ICE)-guided zero-fluoroscopic cryoballoon ablation (CBA) in patients with paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Patients (n=100) undergoing de novo CBA for paroxysmal AF were randomly assigned (1:1) to zero-fluoroscopic (Zero-X) and conventional fluoroscopy groups.

Radiation exposure, procedural time, acute and long term outcome were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing de novo CBA for symptomatic paroxysmal atrial fibrillation

Exclusion Criteria:

* age < 18 years
* history of AF ablation or cardiac surgery
* contraindication to oral anticoagulants
* presence of intracardiac thrombus or significant coronary artery disease on cardiac computed tomography prior to the procedure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Radiation exposure time | 1 day
  comparison of radiation exposure time between the two groups
Radiation exposure dose | 1 day
  comparison of radiation exposure dose between the two groups
acute success rate | 1 day
  successful rate of pulmonary vein isolation
Recurrence rate of atrial tachyarrhythmias | 3 months
  long term outcome : Recurrence rate of atrial tachyarrhythmias 3 months after the procedure

SECONDARY OUTCOMES:
Procedure time | 1 day
  Procedure time between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Hong Euy Lim, MD, Study Chair — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang, South Korea